CLINICAL TRIAL: NCT05791084
Title: Supporting Women With Left Sided Breast Cancer to Practice Deep Inspiration Breath Hold (DIBH) at Home Before Radiation Therapy Treatment
Brief Title: Supporting Women With Breast Cancer to Practice DIBH at Home Before Radiation Therapy
Acronym: DIBHApp
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonkoping University (Other)
Responsible Party: Principal Investigator, Maria Brovall, associated professor, Jonkoping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-04031
Record Dates: First submitted 2023-02-22; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Health Literacy; Distress, Emotional; Preparedness; Mobile Application
Keywords: DIBH; RCT; radiotherapy; mobile application; distress

STUDY DESIGN:
Intervention Model Description: RCT with an intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A=Control group who receives customary information prior to RT with DIBH. (No Intervention): Usual care and information before start of radiotherapy with DIBH.
- B=Intervention group usual care and the DIBH-App to practice at-home before RT with DIBH. (Experimental): Usual care and information and a mobile application with breathing instructions and a sensor to attach around the chest. To be able to train at home before radiotherapy with DIBH starts.
  Interventions: Other: mobile application with breathing instructions and a sensor to attach around the chest. To be able to train at home before radiotherapy with DIBH starts.

INTERVENTIONS:
Other: mobile application with breathing instructions and a sensor to attach around the chest. To be able to train at home before radiotherapy with DIBH starts. — The DIBH-App consists of 1) a mobile application that patients download to their own smart mobile phone, and 2) associated stretch-sensors that are attached around the chest and connected to the mobile phone via Bluetooth. Visually, the graphics is similar to the software used for DIBH in the RT department. Coaching takes place through instructional videos, text, and audio recordings (Image 2). The following information will be recorded and stored: date and time of practice, outcome of each session (including sensor data and calibration parameters), and user behavior within the application (such as screen visits, FAQ sections viewed, and key button presses).
  Arms: B=Intervention group usual care and the DIBH-App to practice at-home before RT with DIBH.

SUMMARY:
To examine the effect of a preparatory digital tool including a new instruction for deep inspiration breath hold (DIBH), before start of radiation therapy in women diagnosed with left sided breast cancer, compared with usual care.

DETAILED DESCRIPTION:
The following questions will be posted:

* Are there any differences in levels of distress (primary outcome) between the control and intervention group at baseline and over time?
* Are there any differences in preparedness for RT (secondary outcomes) between the control and intervention group at baseline and over time?
* Are there any correlations between Health Literacy (HL) levels (secondary outcome) and levels of distress (primary outcome) in the control and intervention group?
* Are there any differences in objective clinical variables (chest mobility and respiratory movements and planned absorbed dose to the heart) between the control and intervention group before and after the intervention (baseline and at planning CT)?
* Which patterns of practice and use of the application (when, how, how often and for how long) can be discerned from the intervention group?
* Are there any correlations between different levels of practice and use of the digital tool and primary and secondary outcomes?
* How do patients in the different groups (control and intervention group) describe their experience of care and information process during RT with DIBH?
* Are there differences regarding health economic variables in terms of costs and health care usage (e.g., estimated time for planning and conducting computed tomography (CT), number of scheduled CT examinations) and patient effects (e.g. co-morbidities (heart related), sick leave, and quality-adjusted life year (QALYs) between patients in control- or interventions group?
* Are there any differences regarding effects on environmental aspects and costs in the different groups (control and intervention)?

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the study:

* patients > 18 years of age
* with a left-sided breast cancer diagnosis or DCIS
* who are to receive RT with DIBH technology
* with curative intention
* preparatory CT visit minimum 7 days to a maximum of 4 weeks
* able to speak and understand good enough Swedish to be able to assimilate content in the mobile app and answer surveys and interview questions
* have access to a smart mobile phone.

Exclusion Criteria:

* patients receiving palliative RT or neoadjuvant chemotherap
* Planning CT starting < 7 days
* people with some form of orthopedic, rheumatological or neurological injury or disease that limits the possibility of carrying out the intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Distress (DIS-A) | Time 1, baseline at randomisation/inclusion
  The Distress Thermometer (DT) was developed as a simple tool to effectively screen for symptoms of distress. The instrument is a self-reported tool using a 0-to-10 rating scale, where 0 is no distress and 10 the worst distress.
Distress (DIS-A) | time 2, at CT-planning visit one week
  The Distress Thermometer (DT) was developed as a simple tool to effectively screen for symptoms of distress. The instrument is a self-reported tool using a 0-to-10 rating scale, where 0 is no distress and 10 the worst distress.
Distress (DIS-A) | time 3, 3 weeks post RT
  The Distress Thermometer (DT) was developed as a simple tool to effectively screen for symptoms of distress. The instrument is a self-reported tool using a 0-to-10 rating scale, where 0 is no distress and 10 the worst distress.
Distress (DIS-A) | time 4, 6 month post RT
  The Distress Thermometer (DT) was developed as a simple tool to effectively screen for symptoms of distress. The instrument is a self-reported tool using a 0-to-10 rating scale, where 0 is no distress and 10 the worst distress.
Distress (DIS-A) | time 5, 5 years after RT
  The Distress Thermometer (DT) was developed as a simple tool to effectively screen for symptoms of distress. The instrument is a self-reported tool using a 0-to-10 rating scale, where 0 is no distress and 10 the worst distress.

SECONDARY OUTCOMES:
HRQoL and Health economic (EQ-5D-5L) | at baseline when inclusion/randomisation
  Health economic measured with EQ-5D-5L a health-related quality of life instrument used to calculate quality-adjusted life years (QALY) . Its design accounts for the need for a direct link between the measurement and valuation of health, whereby every health state that patients might report on the EQ-5D-5L instrument can be summarised by a single value. In order to be used in the calculation of quality-adjusted life years (QALYs; a metric used in cost-utility anal-ysis that combines survival and HRQL), these values need to summarise how good or bad each health state is on a scale anchored at 1 (full health) and 0 (a state equivalent to dead). Values less than 0 represent health states considered to be or modelled as worse than dead.
HRQoL and Health economic (EQ-5D-5L) | 5 years post RT
  Health economic measured with EQ-5D-5L a health-related quality of life instrument used to calculate quality-adjusted life years (QALY) . Its design accounts for the need for a direct link between the measurement and valuation of health, whereby every health state that patients might report on the EQ-5D-5L instrument can be summarised by a single value. In order to be used in the calculation of quality-adjusted life years (QALYs; a metric used in cost-utility anal-ysis that combines survival and HRQL), these values need to summarise how good or bad each health state is on a scale anchored at 1 (full health) and 0 (a state equivalent to dead). Values less than 0 represent health states considered to be or modelled as worse than dead.
e-HL (eHLQ) | at baseline when inclusion/randomisation
  eHealth Literacy Questionnaire-Swedish version, aims to measure a broad range of literacy skills, which could make it useful in assessing the effects of strategies for delivering online information and applications. eHEALS is an 8-item instrument with each item scored on a 5-point Likert scale.Each item is rated on a 5-point. Likert scale, ranging from 1 = strongly disagree to 5 = strongly agree.
Communicative, critical and functional HL | at baseline when inclusion/randomisation
  consists of 14 statements with 4 points Likert scales (1-4). The statements ask how often (never to often) patients have trouble with reading or understanding leaflets from healthcare providers/hospital or pharmacy (functional health literacy; 5 items), have difficulty (easy to rather difficult) performing certain actions in relation to health information (communicative (5 items) and critical (4 items) health literacy).
Preparedness(PCSQ-24) | at CT planning visit, one week
  Modified version of the Preparedness for Colorectal Cancer Surgery Questionnaire, with 28 items measuring preparedness for surgery was developed covering four domains.All items were rated on a Likert-type scale with the following translated response options: Strongly agree, Agree somewhat, Disagree somewhat, and Totally disagree (with corresponding values ranging from 4 to 1)
The Radiotherapy Experience Questionnaire, Swedish modified version | 3 weeks post RT
  The Radiotherapy Experience Questionnaire (RTEQ) with 23 items. This instrument assesses the patient's experiences of the external RT procedure and includes psychological stress, physical discomfort and coping during the external RT procedure.t Likert-type scale for response options, which ranged from 1 = I strongly agree to 6 = I strongly disagree

OTHER OUTCOMES:
Logged data from the CT machine | at Ct planning visit, one week
  will be collected at all treatment occasions on all included patients. Estimation of time for planning CT (min)
Logged data from the CT machine | at Ct planning visit, one week
  number of correct and failed breathing attempts that the patient needs for approved CT. (nr of CT)
Data from the journal | at Ct planning visit, one week
  Data from the journal on all included patients, looking at extra visits for making planning CT.
Logged data from the RT machine | at Ct planning visit, one week
  Logged data from radiation treatment devices (linear accelerators) will be collected at all treatment occasions on all included patients. Estimation of time on RT
Logged data from the CT machine | 3 weeks post RT
  will be collected at all treatment occasions on all included patients. Estimation of time on planning CT (min)
Logged data from the CT machine | 3 weeks post RT
  number of CT images,
Logged data from the journal | 3 weeks post RT
  Logged data from the journal will be collected on all treatment occasions on all included patients. and extra visits during the treatment period and after.
Logged data from RT machine | 3 weeks post RT
  Logged data from the radiation treatment devices (linear accelerators) will be collected at all treatment occasions on all included patients. Estimation of time on RT on each occasion.
Measurement of chest mobility | at baseline when inclusion/randomisation
  Respiratory Objective Measurements. Thorax extension: chest mobility will be measured with a measuring tape, during maximum breathing movements, with the addition of voluntary movements of the chest (the measurement is in centimeters and millimeters)
Measurement of chest mobility | at planning CT, one week
  Respiratory Objective Measurements. Thorax extension: chest mobility will be measured with a measuring tape, during maximum breathing movements, with the addition of voluntary movements of the chest(the measurement is in centimeters and millimeters)
RMMI test | at planning CT visit, one week
  Respiratory movements will be measured on ten patients in the pilot-test, from group B with the Respiratory Movement Measuring Instrument (RMMI) (ReMo Inc. Keldnaholt, Reykjavik, Iceland). The measurement will be performed during maximum breathing movements and is measured bilaterally in the upper and lower part of the thorax and the abdomen. The measurement will be performed by a physiotherapist in the project. The test will evaluate if the measurement with logged data in the app and the respiratory objective measurements are reliable measurements. If not, this measurement will be done to patients in the group B in the RCT study to evaluate the effect.
Planned and given absorbed RT dose to the heart during RT | baseline at inclusion /randomisation
  Given and planned RT-heart dose will be obtained from the journal. Note possibly heart or lung diseases
Planned and given absorbed RT dose to the heart during RT | 5 years post RT
  Given and planned RT-heart dose will be obtained from the journal, 5 years after RT. Note possibly heart or lung diseases
Demographic information. Modified version of The self-administrated comorbidity, The Self-Administered Comorbidity | baseline at inclusion/randomisation
  Modified version of The Self-Administered Comorbidity. Journal data will be collected. Data will be collected regarding type and dose of chemotherapy for control of e.g., heart toxicity, other diseases, medications, sick-leave.
Demographic information, Modified version of The self-administrated comorbidities, The Self-Administered Comorbidity | 5 years follow up post RT
  Modified version of The Self-Administered Comorbidity. Journal data will be collected. Data will be collected regarding type and dose of chemotherapy for control of e.g., heart toxicity, other diseases, medications, sick-leave.
Training patterns | from baseline at inclusion/randomisation
  Number of times practiced and maximal movement at each training session (min vs max). Logged data from app.
Training patterns | up until the CT planning vistit, one week
  Number of times practiced and maximal movement at each training session (min vs max). Logged data from app.
Environmental effects | 3 weeks post RT
  Modes of travelling, distance to clinic (km) and time spent for RT treatment (min). Questions answered i kilometer per mile, time estimation,type of transportation (car, buss, etc).
Focus group interview | 3 weeks post RT
  The focus group interviews are based on open-ended questions, and they will be asked to describe their experience of the care process in breath-adapted radiation therapy (before, during and after the treatment) and the breathing practice based on their group affiliation. Participants are selected within each group with a view to a spread of age, socio-demographic characteristics, and treatment approach.

CONTACTS AND LOCATIONS:
Overall Officials: maria Brovall, ass prof, Principal Investigator — Jonkoping University